CLINICAL TRIAL: NCT01978613
Title: Investigation on Safety, Tolerability and Pharmacokinetics of Multiple Doses of NNC0113-0987 in an Oral Formulation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9927-4022; 2013-000188-10 (EudraCT Number); U1111-1138-4595 (Other: WHO)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oral B (DC) (Experimental): Escalation design. Planned end dose level is 5 mg alternative dosing condition (fasting for 30 minutes post-dosing)
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral D (Experimental): Escalation design. Planned end dose level is 20 mg standard dosing condition (fasting for 120 minutes post-dosing)
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral C (Experimental): Escalation design. Planned end dose level is 10 mg standard dosing condition (fasting for 120 minutes post-dosing)
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral B (Experimental): Escalation design. Planned end dose level is 5 mg standard dosing condition (fasting for 120 minutes post-dosing)
  Interventions: Drug: NNC0113-0987; Drug: placebo
- Oral A (Experimental): Escalation design. Planned end dose level is 2.5 mg standard dosing condition (fasting for 120 minutes post-dosing)
  Interventions: Drug: NNC0113-0987; Drug: placebo

INTERVENTIONS:
Drug: NNC0113-0987 — Tablets for once-daily oral administration. Multiple doses with sequential dose increments over 10 weeks. The end-dose levels and the dose levels during the escalation regime may be adapted during trial conduct based on safety evaluations.
Drug: placebo — Tablets for one-daily oral administration.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) of multiple doses of NNC0113-0987 in an oral formulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, who is considered to be generally healthy, based on the medical history, physical examination, and the results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator
* Age 18-64 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI): 20.0-29.9 kg/m^2 (both inclusive)

Exclusion Criteria:

* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological,dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Subject with previous gastrointestinal surgery, except subjects that underwent uncomplicated surgical procedures such as appendectomy, hernia surgery, biopsies, as well as colonic and gastric endoscopy
* Use of prescription or non-prescription medicinal products and herbal products (except routine vitamins) within three weeks preceding the dosing period. Occasional use of paracetamol or acetylsalicylic acid is permitted

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events recorded | From the time of first dosing (day 0) and until completion of the post-treatment follow-up visit (day 83-97)

SECONDARY OUTCOMES:
Number of hypoglycaemic episodes | From the time of first dosing (day 0) and until completion of the post-treatment follow-up visit (day 83-97)
Area under the NNC0113-0987 plasma concentration time curve | During a dosing interval (0-24 hours) at steady state (day 67, day 68 and day 69)
Maximum observed NNC0113-0987 plasma concentration | During a dosing interval (0-24 hours) at steady state (day 67, day 68 and day 69)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com